CLINICAL TRIAL: NCT05496673
Title: Meningitis: Burden, Causes, Screening and Prevention in Rural Northern Uganda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Lira University (Other); Fogarty International Center of the National Institute of Health (NIH); Makerere University (Other)
Responsible Party: Principal Investigator, Paul Bohjanen, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00007296; R21TW012439 (NIH)
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Meningitis
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with meningitis or risk factors for meningitis (Experimental): Patients who are assessed at outpatient clinics near Lira, Uganda, Lira Regional Referral Hospital emergency room or are admitted to Lira Regional Referral Hospital with meningitis symptoms (defined as headache or irritability in combination with fever, confusion or Glasgow coma scale (GCS) <14, photophobia, neck pain/stiffness, seizure or bulging fontanel) or are deemed at risk for meningitis will be approached to participate in the study. Experimental molecular diagnostic testing such as cryptococcal antigen lateral flow assay, Pastorex antigen agglutination assay and/or Biofire PCR assay will be performed based on HIV status and a clinical assessment identify infectious agents.
  Interventions: Diagnostic Test: Pastorex Latex Agglutination Test; Diagnostic Test: Biofire PCR for meningitis; Diagnostic Test: Immy CrAg Lateral Flow Assay

INTERVENTIONS:
Diagnostic Test: Pastorex Latex Agglutination Test — Rapid diagnosis of bacterial meningitis
Diagnostic Test: Biofire PCR for meningitis — Rapid diagnosis of multiple forms of meningitis
Diagnostic Test: Immy CrAg Lateral Flow Assay — Rapid diagnosis of cryptococcal meningitis

SUMMARY:
This study will investigate the burden, causes, diagnostics, treatments and preventive measures related to meningitis in northern Uganda. We hypothesize that understanding the burden of meningitis, risk factors, diagnostics, treatments and the preventive measures will provide information regarding the gaps in care that can be addressed in order to improve the continuum of meningitis care. we hypothesize that our data will support the advocacy for the implementation of routine vaccination for the prevention of bacterial meningitis and improving guidelines for Cryptococcal antigen (CrAg) screening for prevention of cryptococcal meningitis, which will save lives in Uganda.

Aim 1: To prospectively collect data on 1100 patients with meningitis and meningitis symptoms who were admitted to Lira Regional Referral Hospital (LRRH) to assess burden, etiologies, pathogenesis, and outcomes of meningitis using modern diagnostic testing not previously available in Uganda.

Aim 2: To perform CrAg screening of 10,000 HIV-positive patients to determine the prevalence of cryptococcal antigenemia (infection) and conduct a case control study to compare risk factors and outcomes among CrAg-positive patients and matched CrAg-negative controls based on age, sex, TB status, ART experience, CD4 count, and viral load.

ELIGIBILITY:
Inclusion Criteria:

* 1100 patients who present with meningitis or meningitis symptoms, regardless of age or vulnerably status are eligible for meningitis testing.
* 10,000 HIV-infected patients presenting to LRRH, LRRH HIV Clinic (LIDC) or nearby outpatient clinics, regardless of age or vulnerability status, are eligible for CrAg screening.

Exclusion Criteria:

* Patients who are found not to have meningitis after initial evaluation, or are found to have other alternative diagnoses that explain their symptoms, will be excluded.
* HIV-negative patients without signs or symptoms of meningitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
number of participants with meningitis who died during hospitalization | duration of hospitalization, approximately 2 weeks
number of participants with meningitis who died during the first 24 months after hospital admission | 24 months
number of participants who were screened using the CrAg diagnostic test who were cryptococcal antigen positive | 2 years

SECONDARY OUTCOMES:
number of participants who develop overt cryptococcal meningitis | 2 years
  Overt cryptococcal meningitis is defined as symptomatic meningitis.
Number of participants with overt cryptococcal meningitis who die | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Lira Regional Referral Hospital, Lira, Uganda

IPD SHARING:
Plan to Share IPD: No